CLINICAL TRIAL: NCT04732052
Title: The Use of Transcranial Direct Current Stimulation (tDCS) to Reduce Impulsivity and Aggression in Adults With Developmental Disabilities: The tDCS-RIADD Randomized Controlled Trial Protocol
Brief Title: The Use of Transcranial Direct Current Stimulation (tDCS) in Adults With Developmental Disabilities
Acronym: tDCS-RIADD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Najat Khalifa (Other)
Responsible Party: Sponsor-Investigator, Dr. Najat Khalifa, Principle Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSIY-688-20
Record Dates: First submitted 2020-11-27; First posted 2021-02-01 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Aggression
MeSH Terms: conditions — Aggression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tDCS (Active Comparator): Transcranial Direct Current Stimulation: Soterix tDCS kit will be used to deliver the stimulation using two sponge electrodes soaked in a saline solution. The stimulation montage will comprise of left anodal Dorsal Lateral Prefrontal cortex (DLPFC) stimulation. The anodal electrode will be placed over the area corresponding to the left DLPFC (F5 of the EEG10-20 international system) and the reference (cathodal) electrode over the right supraorbital ridge. The active stimulation condition will use a constant current of 2mA, delivered via gradual increase and decrease over 10 seconds at the onset and offset of stimulation (current ramps), respectively. The duration a single tDCS session will be 20 minutes.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham tDCS (Sham Comparator): Sham Transcranial Direct Current Stimulation: Soterix tDCS kit will be used to deliver the sham stimulation using two sponge electrodes soaked in a saline solution. The sham stimulation montage will comprise of left anodal Dorsal Lateral Prefrontal cortex (DLPFC) stimulation for 10s only. The anodal electrode will be placed over the area corresponding to the left DLPFC (F5 of the EEG10-20 international system) and the reference (cathodal) electrode over the right supraorbital ridge. The sham tDCS is identical to the active tDCS except that the current will be delivered only in the first 10 seconds, after which the stimulation will cease but with the electrodes still in place throughout the session. The duration of each sham tDCS session will be 20 minutes.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — non-invasive brain stimulator

SUMMARY:
Aggressive behaviours are highly prevalent among people with developmental disabilities, both in community and inpatient or residential settings, with adverse consequences for the individuals involved and others. Some predictive factors, particularly impulsivity, are dynamic with neurobiological underpinnings, and as such amenable to change or neuromodulation using non-invasive brain stimulation techniques. With this in mind, we designed an experimental protocol to determine the efficacy of transcranial Direct Current Stimulation (tDCS) as a non-invasive brain stimulation technique to reduce impulsivity and aggression associated with developmental disability.

DETAILED DESCRIPTION:
This study aims to assess the efficacy of anodal tDCS in modulating Rapid Response Impulsivity (RRI) and reducing incidents of aggression in people with developmental disabilities is residential or hospital settings. Using a single blind, parallel arms, randomized controlled trial design, adults (n=60) aged 18 to 65 with developmental disabilities, who have a history of impulsivity leading to aggression, will be randomised to receive either repetitive anodal or sham tDCS. Enrolled participants will receive either three treatment sessions of tDCS or sham tDCS. Behavioural and impulsivity will be measured before and immediately after treatment, one week, and one month after treatment end. Data will be analysed in SPSS using repeated measures ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-64 years
* Diagnosis of a developmental disability
* History of one or more incidents of aggression in the last month
* Consent to participate in the trial by the individual or their Substitute Decision Maker

Exclusion Criteria:

* History of epilepsy or seizures
* History of acquired brain injury
* Having metal in the brain/skull, e.g. splinters, fragments or clips
* Having a cochlear implant
* Having an implanted neuro-stimulator (e.g. direct brain stimulation, epidural/subdural stimulation, vagal nerve stimulation)
* History of brain surgery of procedure
* History of severe adverse reaction to tDCS
* Having a cardiac pacemaker or intracardiac lines
* Current alcohol or drug misuse
* Having a sensitive scalp

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Aggression | change from baseline one week and one month after the third tDCS session
  To determine the effect of tDCS treatment on aggressive symptoms measured by The Modified Overt Aggression Scale (MOAS); Total weighted scores range from 0-40, with a higher score indicating more aggressive behavior.

SECONDARY OUTCOMES:
Maladaptive behaviors | change from baseline one week and one month after the third tDCS session
  Behavior Problems Inventory (BPI); The total frequency scores range from 0-120 and severity of self-injurious behaviour and aggression subscales from 18-54, with higher scores indicating higher frequency and severity
Intervention side effects | Up to 72hrs after the first, second, and third active or sham tDCS treatments.
  Tracking potential side effects of tDCS/sham treatments using tDCS adverse effects questionnaire.
Trait Impulsivity | Baseline
  Barratt Impulsiveness Scale-11 (BIS-11); The total scores range from 30 - 120, with higher scores indicating higher impulsivity.
Impulsivity | change from baseline and the same day after the third tDCS sessions
  To determine the effects of tDCS treatment on symptoms of impulsivity measured by the Stop Signals Task (SST)
Treatment Acceptability | Up to 72hrs after the third active or sham tDCS treatments.
  Total scores on the tDCS Treatment Acceptability Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Ayub, MD, Study Chair — Queen's University
Locations (1):
- Providence Care Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD including all IPD that underlie results in publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All IPD will be available at study end (in two years) and be available for five years following study end date.
Access Criteria: Designated study personnel only